CLINICAL TRIAL: NCT01946230
Title: The Study of p62/SQSTM1 as a Malignant Transformation Marker for Oral Potentially Malignant Disorders and a Prognostic Marker for Oral Squamous Cell Carcinoma
Acronym: p62/SQSTM1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201306005RINC
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Oral Potentially Malignant Disorder; Oral Cancer; Malignant Disorder; p62/SQSTM1
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The mortality rate of oral cancer in Taiwan is still high with no decrease. One of the reasons result in these situations is the patent visits hospital for treatment in late stage of oral cancer. Recently, the government makes effort in oral cancer screening to find oral potentially malignant disorders (OPMD) early. However, there is no conscience in treatment strategies of OPMD up to now. In this study, we will set a OPMD data bank, and use the cases to find out the potential biomarker, which is able to predict the oral cancer malignant transformation. Sixty OPMD with oral cancer transformation will be recruited, and 60 OPMD with no oral cancer malignant transformation will also be enrolled as the disease control group. Besides, 20 normal cases and 60 oral cancer cases resulting from previous OPMD will be collected. All those groups will detect the expression of p62/SQSTM1 to investigate the possibility that p62/SQSTM1 as a biomarker to predict the malignant transformation of OPMM, and a guideline to treat or not to treat OPMD.

ELIGIBILITY:
Inclusion Criteria:

Study group was oral precancerous lesions in patients with malignant transformation; control group was generally no precancerous disease and orthodontic surgery volunteer

Exclusion Criteria:

Oral mucosa of subjects is too thin

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctor of Dental Surgery
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The study of p62/SQSTM1 as a Malignant Transformation Marker for Oral Potentially Malignant Disorders and a Prognostic Marker for Oral Squamous Cell Carcinoma | two year

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hsin Ming, PHD, Principal Investigator — National Taiwan University Hospital